CLINICAL TRIAL: NCT06004778
Title: Lecturer (Academician at University)
Brief Title: The Effect of Motivational Support Program Applied to Adolescents on Sleep Quality and Academic Achievement
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Demet Sokun Ayaz, lecturer, Istanbul University - Cerrahpasa
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: Demet Sokun Ayaz
Record Dates: First submitted 2023-07-20; First posted 2023-08-22 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: High School 11th Grade Students; Absence of Any Language, Hearing, Mental or Psychological Disability; Turkish Speaking and Understanding; Having a PUKI Index Above 5ı; Absence of Any Chronic Disease; Obtaining Permission From Parents and Students
MeSH Terms: interventions — Training Support

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Motivational Support Program (Experimental): Training booklet will be provided.A total of 5 sessions of sleep training will be given by dividing them into groups of 30 minutes, 3 days a week for 2 weeks.Individual motivational interviews will be held with students and reminder messages will be sent twice a week.
  Interventions: Behavioral: Motivational Support Program
- educational support (Active Comparator): Training booklet will be provided. A total of 5 sessions of sleep training will be given by dividing them into groups of 30 minutes, 3 days a week for 2 weeks.
  Interventions: Behavioral: Educational support

INTERVENTIONS:
Behavioral: Motivational Support Program — In studies conducted on adolescents with poor sleep quality, no study using motivational interviewing technique was found.
  Arms: Motivational Support Program
Behavioral: Educational support — educational support
  Arms: educational support

SUMMARY:
It was planned as a randomized controlled experimental study with a single-blind technique, pretest-posttest control group and repetitive measurements, in order to determine the effect of motivational support program applied to adolescents and education on sleep quality.

ELIGIBILITY:
Inclusion Criteria:

* No language disorders
* No hearing disorders
* No mental disorders
* Bad sleep quality
* No chronic disease

Exclusion Criteria:

* Sleeping pill
* Psychiatric illness

Ages: 16 Years to 17 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 84 (Estimated)
Dates: Start 2023-09-13 (Estimated); Primary Completion 2024-01-19 (Estimated); Study Completion 2024-01-19 (Estimated)

PRIMARY OUTCOMES:
Sleep quality Score | up to 2 months (1 OCTOBER 2023-30 NOVEMBER 2023)
  Adolescents receiving motivational support programs have higher average sleep quality scores.

SECONDARY OUTCOMES:
Academic Achievement Score | up to 2 months (1 OCTOBER 2023-30 NOVEMBER 2023)
  Adolescents receiving motivational support program had higher academic achievement averages.

CONTACTS AND LOCATIONS:
Locations (1):
- Demet Sökün Ayaz, Istanbul, Turkey (Türkiye)